CLINICAL TRIAL: NCT01878032
Title: Color Vision as an Outcome Measure for Clinical Trials of Inherited Retinal Degenerations
Brief Title: Color Vision as a Measure for Inherited Retinal Diseases
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130154; 13-EI-0154
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-04-14

CONDITIONS: Healthy Volunteer; Retinal Disease; Inherited Retinal Degeneration
Keywords: Retinal Disease; Inherited Retinal Degeneration
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- The purpose of this study is to find out whether color vision measured with the Cambridge Color Test is a good way to examine the severity of inherited retinal diseases (IRDs). IRDs are a major cause of vision loss worldwide, but very little is known about how the diseases affect color vision over time. This study will tell us if color vision may be used to track changes in inherited retinal diseases over time.

Objectives:

- To improve understanding of color vision as a way to measure changes in inherited retinal diseases.

Eligibility:

* People 5 years of age or older who have an IRD.
* Healthy volunteers at least 5 years of age.

Design:

* Participants will make at least one visit to the National Eye Institute clinic. If they sign up for more tests, they may have up to three visits to the NEI clinic.
* Participants will be asked questions about their medical and eye history.
* Participants will be given an eye exam, including eye drops to dilate their pupils. They will take the Cambridge Color Test, which includes looking at a monitor and pressing a button, and arranging colored circles. Several other tests may be offered, but participants can decline to take them.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
Objective: The aims of this study are to 1) examine the sensitivity of the Cambridge Color Test (CCT) and the low vision CCT (LvCCT) to the severity of retinal disease in inherited retinal degeneration (IRD) by comparing color vision status with changes in photoreceptor structure and function, 2) examine the effects of eccentric fixation and reduction in visual acuity on color discrimination thresholds obtained with the CCT and LvCCT, and 3) establish normal ranges for the CCT and the LvCCT and determine the intra-session and inter-session variabilities for these tests.

Study Population: Up to 59 healthy volunteers and 144 IRD participants age 5 or older will be enrolled in this study.

Design: This study will be comprised of three related projects. For Aim 1, color discrimination thresholds (CCT and LvCCT) and assessments of retinal structure (imaging) and function (perimetry/microperimetry and electroretinogram) will be measured in 144 IRD participants with varying retinal phenotypes and visual acuities. IRD participants will be divided into four major categories: 1) cone & cone-rod dystrophies, 2) rod-cone dystrophies, 3) inherited maculopathies, and 4) inherited retinal dysfunction syndromes. The fourth category will be used for IRDs that do not match the description for categories 1-3 (i.e., x-linked retinoschisis, congenital stationary night blindness). Degree of severity of retinal dysfunction in IRD participants will be determined relative to the normal ranges obtained from the healthy volunteers (see Aim 3a below). For Aim 2 color discrimination thresholds (CCT and LvCCT) will be measured in one eye from 12 healthy volunteers in order to examine the effects of eccentric fixation and reduced visual acuity on color thresholds independent of retinal pathology. Between one and three study visits will be required for this aim. Aim 3 will be comprised of two parts. For Aim 3a, color thresholds will be collected from both eyes (for intraocular variability) of 35 healthy volunteers age 5 or older. For Aim 3B, color discrimination thresholds (CCT and LvCCT) will measured from 12 healthy volunteers twice in one session and then again at a second visit occurring within two months of the initial visit to determine intra-session and inter-session variability.

Outcome Measures: For both the CCT and LvCCT, an overall quantitative measure of color vision will be obtained from the calculation of achromatic area. The sensitivity of CCT and LvCCT will be examined by comparing achromatic area for IRD participants with varying levels of phenotype severity defined by measures of retinal structure and function. Secondary outcomes for this study include: 1) evaluation of sensitivity of the CCT and LvCCT to disease severity,

2) evaluation of the effects of decreased visual acuity and eccentricity on color discrimination thresholds (CCT and LvCCT), 3) establishment of the normal range of color discrimination thresholds (CCT and LvCCT) as a function of age, and 4) determination of intra- and inter-session variabilities of the two tests.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participants must be 5 years of age or older.
  2. Participant (or legal guardian) must understand and sign the protocol s informed consent document.
  3. Participant must be able to cooperate with the testing required for this study.
  4. Participant s eyes must have clarity of ocular media and degree of pupil dilation sufficient to permit adequate fundus photography.
  5. For IRD Participants only:

     1. Participant must have IRD, defined as evidence of retinal rod- and cone-mediated

        dysfunction and degeneration established by standard clinical methods including field tests, ERG, and imaging.
     2. Participant must have a measurable visual acuity.
  6. For Healthy Volunteers only:

     1. Participant must have visual acuity of 20/20 or better.

EXCLUSION CRITERIA:

1. Participant is taking medications known to alter color vision, such as hydroxychloroquine (Plaquenil ), sildenafil (Viagra ), ethambutol, chloroquine amiodarone, and pamidronate disodium.
2. Participant has another ocular disease that may confound the study results, such as diabetic retinopathy, vascular occlusions, retinopathy related to drug toxicity, optic neuropathy, or central serous chorioretinopathy.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-06-03; Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
For both the CCT and LvCCT, a quantitative measure of color vision will be obtained from the calculation of achromatic area. | Ongoing

SECONDARY OUTCOMES:
Determination of variabilities of the two tests | Ongoing
Establishment of the normal range of color discrimination thresholds | Ongoing
Evaluation of effects of disease on color discrimination thresholds | Ongoing
Evaluation of sensitivity of the CCT and LVCCT | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Brett G Jeffrey, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jacobson SG, Cideciyan AV, Ratnakaram R, Heon E, Schwartz SB, Roman AJ, Peden MC, Aleman TS, Boye SL, Sumaroka A, Conlon TJ, Calcedo R, Pang JJ, Erger KE, Olivares MB, Mullins CL, Swider M, Kaushal S, Feuer WJ, Iannaccone A, Fishman GA, Stone EM, Byrne BJ, Hauswirth WW. Gene therapy for leber congenital amaurosis caused by RPE65 mutations: safety and efficacy in 15 children and adults followed up to 3 years. Arch Ophthalmol. 2012 Jan;130(1):9-24. doi: 10.1001/archophthalmol.2011.298. Epub 2011 Sep 12. PMID 21911650
- [Background] Schwartz SD, Hubschman JP, Heilwell G, Franco-Cardenas V, Pan CK, Ostrick RM, Mickunas E, Gay R, Klimanskaya I, Lanza R. Embryonic stem cell trials for macular degeneration: a preliminary report. Lancet. 2012 Feb 25;379(9817):713-20. doi: 10.1016/S0140-6736(12)60028-2. Epub 2012 Jan 24. PMID 22281388
- [Background] Birch DG. A randomized placebo-controlled clinical trial of docosahexaenoic acid (DHA) supplementation for X-linked retinitis pigmentosa. Retina. 2005 Dec;25(8 Suppl):S52-S54. doi: 10.1097/00006982-200512001-00023. No abstract available. PMID 16374336